CLINICAL TRIAL: NCT01740219
Title: Promoting the Utilization of Cancer Early Detection Methods Among Latinos in Church: a Faith-based Approach
Brief Title: Promoting Organizational Capacity to Implement Cancer Control Programs Among Latino Churches
Acronym: CRUZA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Jennifer Allen, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19674
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Cancer
Keywords: Health promotion; Religion and medicine; Hispanic Americans; Randomized controlled trial; Program evaluation; Neoplasms/prevention & control; Mass screening; Female; Male; Preventive Health Services/methods; Adult; Organizations
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capacity Enhancement (Experimental)
  Interventions: Behavioral: Capacity Enhancement
- Standard Dissemination (Active Comparator)
  Interventions: Behavioral: Standard Dissemination

INTERVENTIONS:
Behavioral: Capacity Enhancement — Churches in the Capacity Enhancement intervention will be invited to work with CRUZA staff over the course of a three month intervention to implement health promotion activities in their church and participate in capacity-building educational workshops. Participants may also receive technical assistance from Health Educators in order to implement their cancer education activities.
  Arms: Capacity Enhancement
Behavioral: Standard Dissemination — Churches in the Standard Dissemination arm will receive program materials with information about cancer prevention/early detection and health resources.
  Arms: Standard Dissemination

SUMMARY:
This research study aims to develop an organizational-level intervention to enable communities to adopt, adapt, implement and sustain evidence-based interventions (EBIs) to address cancer disparities among Latinos. The investigators partner with faith-based organizations, since they play a highly prominent role in Latino community life. This three-phase study will: (1) improve understanding of the organizational infrastructure, skills and resources required by Latino churches to implement EBIs for cancer control, (2) develop a capacity-building intervention; and (3) test the intervention's effectiveness in a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Parishes eligible for the Randomized trial are those that are: Roman Catholic, located in Massachusetts, offer religious services in Spanish, and have taken part in the organizational survey.

Exclusion Criteria:

* Not Roman Catholic, not located in Massachusetts, don't offer religious services in Spanish, and have not participated in the organizational survey.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Implementation | 3-months
  Number and types of interventions offered

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Allen, ScD, Principal Investigator — Dana-Farber Cancer Institute; Maria Idali Torres, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (3):
- United States (3):
  - University of Massachusetts Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Tufts University, Medford, Massachusetts

REFERENCES:
- [Derived] Allen JD, Shelton RC, Kephart L, Jandorf L, Folta SC, Knott CL. Organizational characteristics conducive to the implementation of health programs among Latino churches. Implement Sci Commun. 2020 Jul 6;1:62. doi: 10.1186/s43058-020-00052-2. eCollection 2020. PMID 32885217
- [Derived] Allen JD, Shelton RC, Kephart L, Tom LS, Leyva B, Ospino H, Cuevas AG. Examining the external validity of the CRUZA study, a randomized trial to promote implementation of evidence-based cancer control programs by faith-based organizations. Transl Behav Med. 2020 Feb 3;10(1):213-222. doi: 10.1093/tbm/iby099. PMID 30496532
- [Derived] Allen JD, Torres MI, Tom LS, Leyva B, Galeas AV, Ospino H. Dissemination of evidence-based cancer control interventions among Catholic faith-based organizations: results from the CRUZA randomized trial. Implement Sci. 2016 May 18;11(1):74. doi: 10.1186/s13012-016-0430-6. PMID 27193768